CLINICAL TRIAL: NCT03368586
Title: Accuracy, Satisfaction and Usability of a Flash Glucose Monitoring System Among Children and Adolescents Attending a Diabetes Camp
Brief Title: Accuracy, Satisfaction and Usability of a FGM System Among Children and Adolescents Attending a Diabetes Summer Camp
Status: Completed | Type: Observational
Sponsor: University of Lausanne Hospitals (Other)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Michael Hauschild, Dr., University of Lausanne Hospitals
Other Study IDs: CER-VD 2016-00852
Record Dates: First submitted 2017-11-24; First posted 2017-12-11 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Flash Glucose Monitoring; Children; Adolescents
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Flash Glucose Monitoring — The camp comprised a structured daily routine with five fixed meals: breakfast, lunch, afternoon snack, dinner and evening snack. Capillary blood glucose (BG) values were measured in parallel with unmasked Flash Glucose (FG) measurements using the FGM reader's built-in glucometer at breakfast, lunch and dinner. Additional measurements were taken before snacks, between the meals or overnight and BG was measured only in cases of low (<4.0 mmol/L) or high (>15.0 mmol/L) FG values or when symptoms were discordant with sensor readings. Sensor-related issues were documented and a questionnaire assessing satisfaction and usability of the FGM was completed by patients and caregivers at study completion.

SUMMARY:
The aim of this study was to assess accuracy, satisfaction and usability of the FGM among children and adolescents with T1DM. The primary outcome was to assess the accuracy of the FGM system. Secondary outcomes included satisfaction and usability of the device as well as assessment of sensor-related issues.

DETAILED DESCRIPTION:
The aim of this study was to assess the accuracy, satisfaction and usability of a Flash Glucose Monitoring system (FGM) in children and adolescents with type 1 diabetes mellitus (T1DM) and attending a 1-week diabetes summer camp, supervised by a multidisciplinary team of health care providers. The camp comprised a structured daily routine with five fixed meals: breakfast, lunch, afternoon snack, dinner and evening snack. Capillary blood glucose (BG) values were measured in parallel with unmasked Flash Glucose measurements (FGM) using the FGM reader's built-in glucometer at breakfast, lunch and dinner. Additional measurements were taken before snacks, between the meals or overnight and BG was measured only in cases of low (<4.0 mmol/L) or high (>15.0 mmol/L) FGM values or when symptoms were discordant with sensor readings. Sensor-related issues were documented and a questionnaire assessing satisfaction and usability of the FGM was completed by patients and caregivers at study completion.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus, children and adolescents participating at the diabetes summer camp.

Exclusion Criteria:

* Acute health condition (infectious disease), known allergy to medical adhesives or with a skin condition (e.g. atopic dermatitis)).

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents, aged 6-18 years old, with type 1 diabetes mellitus, participating at the diabetes summer camp.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2016-07-02 (Actual); Primary Completion 2016-07-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
FGM accuracy | through study completion, 1 week
  Accuracy of FGM values versus reference blood glucose values (Consensus Error Grid (CEG) analysis and calculation of the Mean Absolute Relative Difference (MARD))

SECONDARY OUTCOMES:
Participants satisfaction with the FGM system | At last camp day
  Participants satisfaction (Questionnaire,%)
Caregivers satisfaction with the FGM system | At last camp day
  Caregivers satisfaction (Questionnaire,%)
Sensor related-issues | Through study completion, 1 week
  Sensor related-issues will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hauschild, MD, Principal Investigator — Lausanne University Hospitals

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and informed consent form will be publicly available. Individual participant data (IPD) collected in this study, including participants individual data, cannot be shared.
Supporting Information: Study Protocol, ICF
Time Frame: study end
Access Criteria: not yet defined